CLINICAL TRIAL: NCT01422811
Title: Unnecessary, Avoidable Lengths of Stay: a Strategy for Clinician Empowerment and Effectiveness Evaluation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Principal Investigator, Caterina Caminiti, Dr., Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: aopr-rct-los
Record Dates: First submitted 2011-08-23; First posted 2011-08-24 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Hospitalization; Length of Stay
Keywords: Public health; Policy; Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Multicomponent strategy to reduce avoidable length of stay
- Control (Other): No Intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Multicomponent strategy to reduce avoidable length of stay — The strategy comprises two integrated components:
  1. Distribution of two monthly reports, one consisting in the list of patients who, through data collection performed, are classified to be present on the ward although their clinical status is considered compatible with discharge; the other featuring individual length of stay profiles for each physician operating in the intervention arm (information taken from administrative data), allowing comparisons with the rest of the medical staff;
  2. Audits performed by professionals of each ward of the intervention arm designed to discuss cases judged to be compatible with discharge. The organization of this work are left to the wards, without any interference from the project team.
  Arms: Intervention
Other: No intervention — No interventions (reporting, auditing) are planned; nevertheless control ward physicians know study aims and are informed about their patient's data collection.
  Arms: Control

SUMMARY:
1. Background: In recent years an increasing trend in excessive lengths of stay has been recorded at the Parma University Hospital, compared with regional mean values. Excessive lengths of stay have been demonstrated to constitute not just an economic problem, but also a clinical and public health issue. Since the measures taken at our institution so far have not proven effective, the investigators carried out a literature review, which mostly detected observational studies, restricted to the assessment of the impact of a single intervention.
2. Objectives: This project intends to evaluate the effectiveness of a multifaceted strategy aiming to empower clinicians on the issues associated with excessively long and avoidable hospital stays, and enable them to identify corrective measures (according to the principles of clinical governance).
3. Study design: cluster-randomized, parallel group, open-label, community trial
4. Methods: trained personnel will periodically record causes for excessive lengths of stay in all participating wards using an ad hoc data collection sheet. In the wards randomized to the experimental group, interventions aimed to clinician empowerment - provision of reminders and periodical audits - will be implemented.
5. Expected results: A reduction in the experimental vs. the control arm unnecessary lengths of stay is expected, although the introduced measures will also presumably lead to improvement in the wards where they are not implemented.

ELIGIBILITY:
Inclusion Criteria:

* patients present on the participating wards during one of 12 randomly selected index days (one for each month of data collection)

Exclusion Criteria:

* patients admitted or discharged on the index days
* patients with length of stay (interview date - admission date) > 90 days

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3862 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patient-days compatible with discharge | 12 month period [02/2008 - 02/2009] +1 follow up month [02/2010]

SECONDARY OUTCOMES:
Overall length of stay (in days) | 12 month period [02/2008 - 02/2009]
  Overall length of stay = discharge date - admission date

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Caminiti, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, Italy

REFERENCES:
- [Background] Carey MR, Sheth H, Braithwaite RS. A prospective study of reasons for prolonged hospitalizations on a general medicine teaching service. J Gen Intern Med. 2005 Feb;20(2):108-15. doi: 10.1111/j.1525-1497.2005.40269.x. PMID 15836542
- [Background] Lagoe RJ, Westert GP, Kendrick K, Morreale G, Mnich S. Managing hospital length of stay reduction: a multihospital approach. Health Care Manage Rev. 2005 Apr-Jun;30(2):82-92. doi: 10.1097/00004010-200504000-00002. PMID 15923910
- [Background] Moro ML. Health care-associated infections. Surg Infect (Larchmt). 2006;7 Suppl 2:S21-3. doi: 10.1089/sur.2006.7.s2-21. PMID 16895497
- [Background] Selker HP, Beshansky JR, Pauker SG, Kassirer JP. The epidemiology of delays in a teaching hospital. The development and use of a tool that detects unnecessary hospital days. Med Care. 1989 Feb;27(2):112-29. doi: 10.1097/00005650-198902000-00003. PMID 2918764
- [Background] Setrakian JC, Flegel KM, Hutchinson TA, Charest S, Cote L, Edwardes MD, Corbett IB. A physician-centred intervention to shorten hospital stay: a pilot study. CMAJ. 1999 Jun 15;160(12):1735-7. PMID 10410639
- [Background] Shojania KG, Wald H, Gross R. Understanding medical error and improving patient safety in the inpatient setting. Med Clin North Am. 2002 Jul;86(4):847-67. doi: 10.1016/s0025-7125(02)00016-0. PMID 12365343
- [Background] Meschi T, Fiaccadori E, Cocconi S, Adorni G, Ridolo E, Stefani N, Schianchi T, Novarini A, Spagnoli G, Caminiti C, Pini M, Borghi L. [Analysis of the problem of "difficult hospital discharges" in the University Hospital of Parma]. Ann Ital Med Int. 2004 Apr-Jun;19(2):109-17. Italian. PMID 15317271
- [Derived] Caminiti C, Meschi T, Braglia L, Diodati F, Iezzi E, Marcomini B, Nouvenne A, Palermo E, Prati B, Schianchi T, Borghi L. Reducing unnecessary hospital days to improve quality of care through physician accountability: a cluster randomised trial. BMC Health Serv Res. 2013 Jan 10;13:14. doi: 10.1186/1472-6963-13-14. PMID 23305251
- See also: Study sponsor's website [ita] — http://www.regione.emilia-romagna.it/